**Study Title:** Impulsivity Mediation Using Transcranial Direct Current Stimulation Paired with Acceptance Commitment Therapy as an Adjunctive Therapy for Substance Use Disorder

STUDY00000768

7/19/2022




Consent Version: 06/20/2022

# **Consent to Participate in Research**

Study Title: Impulsivity Mediation Using Transcranial Direct Current Stimulation Paired with Acceptance Commitment Therapy as an Adjunctive Therapy for Substance Use Disorder

Principal Investigator: Allison J. Huff (allison7@arizona.edu)

#### Sponsor and/or Funder

This study is funded through a seed grant from the Department of Family and Community Medicine in the College of Medicine.

# Summary of the research

**This is a consent form for participation in a research study.** Your participation in this research study is voluntary. It contains important information about this study and what to expect if you decide to participate. Please consider the information carefully. Feel free to ask questions before making your decision whether to participate.

The purpose of this study is to determine the impact of tDCS, a non-invasive brain stimulation treatment that uses low amplitude direct electrical currents to stimulate specific parts of the brain. This study will use an investigational device called the tKIWI to deliver tDCS to participants in recovery from a history of substance use disorder (SUD). The tKIWI is a product of a ni2o, inc. tDCS is recognized to be a safe, non-invasive brain stimulation treatment. This treatment has been widely studied for a number of neurodegenerative brain disorders, and literature reports minimal side effects, which may include tingling at the site of the electrode, slight burning upon treatment, itching at the site during the treatment, and redness at the site of the electrode, headache, and discomfort. All of the potential side effects have been reported to be temporary and transient. For example, when tingling and itching occurs, it has been reported to last approximately ten minutes after treatment ends. If there is any redness at the site the electrode is placed, it has been reported to last up to a couple of days due to the increased blood flow to that area during treatment of tDCS.

Participants in this study are required to have a diagnosis of SUD, but not currently be using substances. The overarching goal of this study is to provide personalized treatment for SUD by decreasing impulsivity, a proxy for cravings.

By agreeing to participate in this study, you are agreeing to attend 7 study sessions. During the first visit, you will be asked to complete an interview or form documenting your demographic information and SUD/relapse history. You will then be asked to fill out a 30-question survey to measure of your level of impulsiveness (Barrett Impulsiveness Survey (BIS-11). We will then measure your brain waves using an electroencephalogram (EEG). An EEG is a test that measures electrical activity in the brain using small, electrodes attached to the scalp. Your brain cells communicate via electrical impulses and are active all the time, even during sleep. This activity

HSPP Use Only: Consent form Medical v2022-05-19




Consent Version: 06/20/2022

shows up as wavy lines on an EEG recording. Once we have this initial measurement, you will participate in a guided imagery activity grounded in Acceptance Commitment Therapy (ACT) and we will record your brain waves again with an EEG. This first session may take up to 1.5 hours.

Visits 2-6 will consist of a pre-treatment EEG, a twenty-minute tDCS session, broken in to three different sessions, and a post-treatment session EEG. You will also report any side-effects during each visit by filling out a brief survey. Vitals (heart rate, pulse, blood pressure temperature) will also be taken at the beginning of each session and at the end of each session. Study visits 2-6 could take between 1-1.5 hours.

The final visit will consist of a final EEG, ACT exercise, and BIS-11 survey. This visit will take approximately 1 hour.

## Why is this study being done?

The purpose of this study is to determine the impact of tDCS, a non-invasive brain stimulation treatment that uses low amplitude direct electrical currents to stimulate specific parts of the brain. This study will use an investigational device called the tKIWI to deliver tDCS to participants in recovery from a history of substance use disorder (SUD).

## What will happen if I take part in this study?

Once recruited, you will be randomly placed in one of two groups. One group will receive the tDCS treatment and the other group will receive a placebo tDCS treatment. Each participant has a 50% chance to be in either the treatment group or the nontreatment group. Both the treatment and sham groups will participate in the ACT activity.

Participants in this study are required to have a diagnosis of SUD, but not currently be using substances. The overarching goal of this study is to provide personalized treatment for SUD by decreasing impulsivity, a proxy for cravings.

## How long will I be in this study?

By agreeing to participate in this study, you are agreeing to attend 7 study sessions over approximately a two-week period.

#### How many people will take part in this study?

We are recruiting 30 participants for this single blind clinical trial. A single blind clinical trial means that participants will be randomly selected to one of two groups.

#### What benefits can I expect from being in this study?

If you are in the treatment group, you may reasonably expect a decrease in impulsivity from participation in the study. If you are placed in the nontreatment group, your participation will

HSPP Use Only:

Consent form Medical v2022-05-19




Consent Version: 06/20/2022

be contributing to an innovative and non-invasive, non-habit forming, safe treatment for addictive behaviors. Both groups may receive a benefit from participating in the Acceptance Commitment Therapy guided imagery activity.

#### What risks, side effects or discomforts can I expect from being in the study?

The risk is minimal and any discomfort you may feel should be minor and temporary, as outlined in the Procedures and Protocols section.

## What other choices do I have if I do not take part in this study?

Your participation in this study is voluntary, and you may withdraw at any time without any negative consequences to you or without penalty or loss of benefits to which you are otherwise entitled. If you choose to withdraw, we will use the data we have collected from you up until your date of withdrawal. If you do not want us to use data we have collected from you, please notify us upon your withdrawal. There are no alternative procedures related to this study, other than to not participate.

## When may participation in the study be stopped?

If, at any time and for any reason, you elect to leave the study, you may do so without any repercussions to you. Our preference is for you to notify our research staff via email or telephone if possible so we can appropriately debrief you. We will use the data we have collected up until the point of your study departure unless you request in writing otherwise.

#### What happens if I am injured because I took part in this study?

If you should experience any of the possible side effects indicated above that require attention, please notify the research team immediately, or email the PI, Dr. Allison J. Huff. Because the possible risks to you are minimal and if they occur are expected to be temporary, we do not offer compensation for experiencing one of the more commonly reported side-effects listed under the Procedures and Protocols section. However, general first aid will be available to address any superficial side-effects. We do not provide compensation for the unlikely event of a more serious side effect/injury. Medical care is not available on site or covered through this grant. However, if you suffer an injury from participating in this study, you should seek treatment.

## What are the costs of taking part in this study?

There is no cost to you for participating in this study other than your time. The transcranial direct current stimulation (tKIWI device) and services performed for research only will be provided at no charge to you or your insurance company.

#### Will I be paid for taking part in this study?

You will be compensated a total of \$175 upon completion of the study. You will receive the payments in cash in the amounts outlined herein: \$25 at visit 1; \$50 at visit 4; and \$100 at visit

HSPP Use Only:

Consent form Medical v2022-05-19



#### 

Consent Version: 06/20/2022

7. Compensation for participation in a research study is considered taxable income for you. If your compensation for this research study or a combination of research studies is \$600 or more in a calendar year (January to December), you will receive an IRS Form 1099 to report on your taxes. Please note, if you are an employee of UArizona, any compensation from a research study is considerable taxable income.

For any compensation or reimbursement you receive, we are required to obtain identifiable information such as your name, address, and Social Security number for financial compliance purposes. Identifiable information collected for financial compliance purposes will not be linked to your research data. If you do not want us to collect this information, you can still participate in this study, but you will not be able to receive any payment for your participation.

#### Will my data be stored for future research?

Deidentified raw EEG and tDCS data may be stored for future research and may possibly be used to identify different biomarkers and further train algorithms. The deidentified EEG and tDCS data will be shared with industry partner, ni20, inc., as per our data sharing agreement.

#### Will my data be sold for commercial profits?

Your data will not be sold for commercial profit.

## Will I hear back on any results that directly impact me?

The results of this trial will be submitted for publication in peer reviewed journals, but you will not be notified of results that directly impact you.

#### Will my study-related information be shared, disclosed, and kept confidential?

It is anticipated there will be circumstances where your study related information and data will be released to persons and organizations described in this form. If you sign this form, you are giving permission to the research team to use and/or disclose your data and demographics for this study. Your information may be shared or disclosed with others to conduct the study, to comply with regulations, and to help ensure that the study has been done correctly. These other groups may include:

- Office for Human Research Protections, Food and Drug Administration, or other federal, state, or international regulatory agencies
- The University of Arizona (UA) and the UA Institutional Review Board
- The sponsor and/or funder supporting the study, their agents or study monitors

#### Who can answer my questions about this study?

If at any time you feel you have had a research-related injury, or for questions, concerns, or complaints about the study you may contact Allison J. Huff, DHEd (Principal Investigator).

HSPP Use Only:

Consent form Medical v2022-05-19



Printed name of person obtaining consent


Consent Version: 06/20/2022

Date

For questions about your rights as a participant in this study or to discuss other study-related concerns or complaints with someone who is not part of the research team, you may contact the Human Subjects Protection Program Director at 520-626-8630 or online at https://research.arizona.edu/compliance/human-subjects-protection-program.

| read to me) this form, and I am award<br>dy. I have had the opportunity to ask<br>. I voluntarily agree to participate in t<br>is form. I will be given a signed copy o | questions and have had them his study. I am not giving up |
|---|---|
| Signature of subject | Date |
| h to the participant or the participant'<br>above. There are no blanks in this doc<br>participant or to the participant's repr | cument. A signed copy of this |
| | dy. I have had the opportunity to ask I voluntarily agree to participate in t is form. I will be given a signed copy of Signature of subject h to the participant or the participant above. There are no blanks in this doc |

Signature of person obtaining consent